CLINICAL TRIAL: NCT00453141
Title: Betamethasone Dosing Interval - 12 or 24 Hours?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cooper Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06030
Record Dates: First submitted 2007-03-26; First posted 2007-03-28 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-03

CONDITIONS: Preterm Delivery
Keywords: Betamethasone for preterm labor; Preterm delivery; Infant Respiratory Distress Syndrome
MeSH Terms: conditions — Premature Birth; Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: dosing of Betamethasone

SUMMARY:
The purpose of this study is to determine if there may be a benefit to the newborn if betamethasone is given 12 hours apart instead of 24 hours apart.

DETAILED DESCRIPTION:
Betamethasone is a medicine given to women expected to deliver after 24 but before 34 weeks of pregnancy. It is very advantageous in preventing or decreasing the many problems these small babies may face if born early. Betamethasone makes breathing easier for them, also decreases the chance of them bleeding in the head and makes their chances of survival better. This medicine is used routinely in pregnancy but the best timing between doses in not well established. The 'standard' dosing schedule involves giving 2 injections of 12mg of the medicine 24 hours apart. However, many women deliver before reaching the 24-hour mark, despite the doctors best efforts to try and delay delivery, and therefore miss the opportunity for the 2nd dose.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women expected to deliver preterm (either induced or spontaneously) for any obstetrical or medical indication.
* Gestational age between 23 and 34 weeks gestational age.
* Dating must either be by LMP which is consistent with ultrasound performed at any gestational age, or calculated by a sonogram less than or equal to 23 weeks.

Exclusion Criteria:

* Patients at <23 or >34 weeks gestational age.
* Known drug allergy to betamethasone.
* Given steroid other than betamethasone for lung maturation.
* Any contraindication to steroid therapy.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The diagnosis of RDS is defined as: PaO2 < 50 mm Hg in room air, central cyanosis in room air, or a requirement for supplemental O2 to maintain PaO2 > 50 mm Hg, along with chest xray findings consistent with RDS (per the Vermont Oxford Network) | Until neonatal discharge

SECONDARY OUTCOMES:
Incidence of INH, NEC, BPD, Blindness | until neonatal discharge

CONTACTS AND LOCATIONS:
Overall Officials: Meena Khandelwal, MD, Principal Investigator — The Cooper Health System
Locations (2):
- United States (2):
  - Cooper University Hospital, Camden, New Jersey
  - Atlanticare Regional Medical Center, Pomona, New Jersey

REFERENCES:
- [Background] Liggins GC, Howie RN. A controlled trial of antepartum glucocorticoid treatment for prevention of the respiratory distress syndrome in premature infants. Pediatrics. 1972 Oct;50(4):515-25. No abstract available. PMID 4561295